CLINICAL TRIAL: NCT05102617
Title: Post Market Usability Evaluation Of The PicoSure Pro Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7051-PM01-2021
Record Dates: First submitted 2021-10-25; First posted 2021-11-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Wrinkle; Acne Scars; Benign Epidermal Pigmented Lesions; Benign Dermal Pigmented Lesions; Tattoo Removal
MeSH Terms: interventions — Cosmeceuticals

STUDY DESIGN:
Masking Description: Randomization is not used for determining which arm subjects will participate in, however, it will be used to determine which side of the treatment area will receive which treatment regimen (if in a group receiving split-face treatments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group A: Split-Face Device Only Treatment (Experimental): Subjects will receive a split face treatment with the PicoSure Pro and/or PicoSure devices using different device settings on each half of the face.
  Interventions: Device: PicoSure Pro Device; Device: PicoSure Device
- Group B: Split-Face Treatment with Cosmeceuticals (Experimental): Subjects will receive a full face treatment with the PicoSure Pro or PicoSure device and will use topical cosmeceuticals on only half of their face.
  Interventions: Device: PicoSure Pro Device; Device: PicoSure Device; Drug: Topical Cosmeceuticals
- Group C: Device Only Treatment (Experimental): Subjects will receive treatments with the PicoSure Pro or PicoSure device on multiple areas of the body such as the face, décolletage, back, legs, arms, and hands.
  Interventions: Device: PicoSure Pro Device; Device: PicoSure Device

INTERVENTIONS:
Device: PicoSure Pro Device — This device will be used for up to 4 treatments over the designated areas.
Device: PicoSure Device — This device will be used for up to 4 treatments over the designated areas.
Drug: Topical Cosmeceuticals — Topical cosmeceuticals, such as a hydrating serum or cream, will be applied on the designated area.
  Arms: Group B: Split-Face Treatment with Cosmeceuticals

SUMMARY:
The intended use of the PicoSure and PicoSure Pro devices used in this study is to treat additional patients with the new PicoSure Pro device and collect additional data on the devices.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are a healthy male or female 18 years of age or older. Up to 100 subjects will be enrolled at up to 4 study centers. Subjects will be enrolled into one of the 3 groups; Group A, Group B, or Group C.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 years of age or older.
* Willing to undergo treatments with the PicoSure and PicoPro devices for pigmentary lesions, acne scars, skin revitalization, or tattoo removal.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
* The subject is hypersensitive to light in the near infrared wavelength region.
* The subject takes medication which is known to increase sensitivity to sunlight.
* The subject has seizure disorders triggered by light.
* The subject takes or has taken oral isotretinoin, such as Accutane®, within the last six months.
* The subject has an active localized or systemic infection, or an open wound in area being treated.
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated.
* The subject has common acquired nevi that are predisposed to the development of malignant melanoma.
* The subject has herpes simplex in the area being treated.
* The subject is receiving or has received gold therapy.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months to entering this study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

* Has unprotected sun exposure within four weeks of treatment, including the use of tanning beds or tanning products, such as creams, lotions and sprays may interfere with the laser treatment; Investigator discretion is required to determine feasibility of treatment administration.
* Has a coagulation disorder or is currently using anti-coagulation medications. Anticoagulants may cause excessive bleeding and interfere with posttreatment healing; Investigator discretion is required to determine feasibility of treatment administration for subjects taking anticoagulants.
* Is taking medications that alter the wound-healing response which may interfere with posttreatment healing and may require special precautions to be taken by a treating Investigator.
* Is known to have a history of healing problems or history of keloid formation, Investigator discretion is required to determine the feasibility of treatment administration.
* Has a history of skin cancer or suspicious lesions, Investigator discretion is required to determine feasibility of treatment administration.
* Has had a chemical or mechanical epilation within the last six weeks may interfere with the post treatment healing process; Investigator discretion is required to determine feasibility of treatment administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Grading of Pre-Treatment vs. Follow Up Images | 30 day follow up
  The investigator will grade the improvement they noticed between the baseline image and the follow up image based on the Global Aesthetic Improvement Scale (GAIS), which ranges from 1-5 as follows: Very Much Improved (1), Much Improved (2), Improved (3), No Change (4), Worse (5).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Director of Clinical Research; Sean Doherty, Principal Investigator — Cynosure, Inc.; Emil Tanghetti, Principal Investigator — Center for Dermatology and Laser Surgery
Locations (2):
- United States (2):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Cynosure, Inc., Westford, Massachusetts

IPD SHARING:
Plan to Share IPD: No